CLINICAL TRIAL: NCT02492841
Title: Controlled Clinical Trial of the Effect of Calcium Hydroxide, Mineral Trioxide Aggregate (MTA) and Biodentine (Trademark) as Direct Pulp Capping Materials of Permanent Teeth Affected by Caries, in Children From 7 to 16 Years
Brief Title: Calcium Hydroxide, Mineral Trioxide Aggregate and Biodentine (Trademark) as Direct Pulp Capping of Permanent Teeth
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Dra. Claudia Brizuel, DDS, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RPD-7-16; SA13I20175 (Other Grant/Funding Number: FONIS SA13I20175)
Record Dates: First submitted 2015-05-27; First posted 2015-07-09 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Caries; Dental Pulp Exposure
Keywords: dentin substitute; vital pulp therapy; Biodentine; caries
MeSH Terms: conditions — Dental Pulp Exposure | interventions — mineral trioxide aggregate; Calcium Hydroxide; tricalcium silicate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mineral trioxide aggregate (MTA) (Experimental): Mineral trioxide aggregate Root canal repair material
  Interventions: Drug: Mineral trioxide aggregate
- Calcium hydroxide (Active Comparator): -material for pulp capping
  Interventions: Drug: Calcium hydroxide
- Biodentine (Experimental): Is a calcium-silicate based materia root perforations, apexification, resorptive lesions, and retrograde filling material in endodontic surgery, pulp capping
  Interventions: Drug: Biodentine

INTERVENTIONS:
Drug: Mineral trioxide aggregate — Mineral trioxide aggregate
  Other Names: MTA Pro Root
  Arms: Mineral trioxide aggregate (MTA)
Drug: Calcium hydroxide — Classic calcium hydroxide root canal repair material. Inorganic compound (CA(OH)2. It is the gold standard direct pulp cupping material.
  Other Names: Calcium hydroxide Hertz
  Arms: Calcium hydroxide
Drug: Biodentine — Biodentine (trademark). Septodont. Biodentine root canal repair material. A predose capsule plus five drops of calcium chloride solution.
  Other Names: Active biosilicate. Septodont.
  Arms: Biodentine

SUMMARY:
Background: Dental caries is considered an oral health problem worldwide. In Chile the last national epidemiological study (2007) showed a national prevalence of dental caries in children 6 years (70.3%) and 12 (62.5%). Direct pulp capping is a preventive dental therapy, keeps the vitality of the tooth using some inductive materials mineralized tissue formation.

Objective: The main objective of this study is to evaluate the effectiveness of two innovative direct pulp capping materials; Biodentine compared MTA and calcium hydroxide in the maintenance of pulp vitality in teeth permanent molars.

DETAILED DESCRIPTION:
Methodology: It is a randomized controlled study. groups signed the informed consent for clinical trial patients, a clinical evaluation of 90 permanent molars teeth through endodontic diagnostic tests and radiograph. will be conducted to determine diagnosis. Will be assigned randomly to the type of material to use and direct pulp teeth affected by caries coating is carried out; Patients will not have knowledge of the material to be used in the coating. The patient will be clinically evaluated at 1 week, 3 months and 8 months, and radiographically; at the beginning and end of the study. In each clinical control endodontic diagnostic tests of heat, cold, electric and percussion will be performed. In radiographic controls take a radiograph control with positioner or surveyor at baseline and 8 months, to evaluate the periapical status. Clinical success will consider that tooth in continuous controls and after 8 months presented vitality and radiographic signs of apical image without injury. Failure unresponsive to consider whether susceptibility testing of cold and electricity in more than one control and presents radiographic image with apical lesion.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients
* Patients with at least one full or partial tooth root development
* Clinical examination of the tooth must be selected diagnostic tests that are consistent with reversible pulpitis
* Radiographic examination should show images of normal tissues without signs of internal resorption, the remaining healthy coronary should be sufficient for an indication of direct restoration
* Teeth that have pulp exposure not exceeding 1 mm in size.

Exclusion Criteria:

* Every child with systemic and / or neurological conditions that make it impossible to focus on conventional dental clinic
* Teeth uncontrolled excessive bleeding during communication pulp those aiming or have plans to move during that time period of 8 months .

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Brizuela, Principal Investigator — Universidad de Los Andes
Locations (1):
- Centro de Salud de San Bernardo Universidad de Los Andes, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paranjpe A, Zhang H, Johnson JD. Effects of mineral trioxide aggregate on human dental pulp cells after pulp-capping procedures. J Endod. 2010 Jun;36(6):1042-7. doi: 10.1016/j.joen.2010.02.013. Epub 2010 Mar 15. PMID 20478462
- [Background] Leye Benoist F, Gaye Ndiaye F, Kane AW, Benoist HM, Farge P. Evaluation of mineral trioxide aggregate (MTA) versus calcium hydroxide cement (Dycal((R)) ) in the formation of a dentine bridge: a randomised controlled trial. Int Dent J. 2012 Feb;62(1):33-9. doi: 10.1111/j.1875-595X.2011.00084.x. PMID 22251035
- [Background] Nowicka A, Lipski M, Parafiniuk M, Sporniak-Tutak K, Lichota D, Kosierkiewicz A, Kaczmarek W, Buczkowska-Radlinska J. Response of human dental pulp capped with biodentine and mineral trioxide aggregate. J Endod. 2013 Jun;39(6):743-7. doi: 10.1016/j.joen.2013.01.005. Epub 2013 Apr 10. PMID 23683272

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mineral Trioxide Aggregate (MTA) | Calcium Hydroxide | Biodentine
Started | 56 | 53 | 60
Completed | 22 | 22 | 25
Not Completed | 34 | 31 | 35
Not completed — Lost to Follow-up | 34 | 31 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mineral Trioxide Aggregate (MTA) | Calcium Hydroxide | Biodentine | Total
Number analyzed (Participants) | 56 | 53 | 60 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.51 (2.34) | 11.64 (2.65) | 11.22 (2.34) | 11.44 (2.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 29 | 87
  Male | 27 | 24 | 31 | 82
Tooth [Count of Participants; unit: Participants]
  Maxillary First molar | 16 | 11 | 17 | 44
  Maxillary Second molar | 1 | 0 | 1 | 2
  Mandibular First molar | 32 | 36 | 36 | 104
  Mandibular Second molar | 7 | 6 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Parameters Evaluated After Treatment
Description: vitality test with electric device cold and hot test radiographic evaluation
Time Frame: 3 months, 6 moths and 12 months
Population: Intent a preventive treatment against cavities to avoid endodoncies with different treatments and see which one is more effective after 12 months follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Mineral Trioxide Aggregate (MTA) | Calcium Hydroxide | Biodentine
Number analyzed (Participants) | 22 | 22 | 25
Participants
  Succesfull treatment | 19 | 19 | 25
  Need other treatment | 3 | 3 | 0

2. Secondary Outcome: Number of Participants With Adverse Effects
Description: Name any adverse effects caused by treatment.
Time Frame: 1 week, 3 and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mineral Trioxide Aggregate (MTA) | Calcium Hydroxide | Biodentine
Number analyzed (Participants) | 22 | 22 | 25
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Mineral Trioxide Aggregate (MTA) | Calcium Hydroxide | Biodentine
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/25

LIMITATIONS AND CAVEATS:
The small sample due to inclusion criteria. Lack of collaboration from the primary health providers. And the fact that the oral health seems not to be a priority and people only come when it hurts and it is too late for prevention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No